CLINICAL TRIAL: NCT01117649
Title: Prospective, Controlled, Double-blind, Randomized Multi-centric Study on the Efficacy and Safety of a Target Controlled PVR Therapy With a Hyperoncotic Balanced Hydroxyethyl Starch (HES) Solution Versus an Isooncotic Balanced HES Solution Compared to a Balanced Electrolyte Solution in Elective Surgery
Brief Title: Plasma Volume Replacement (PVR) Therapy With Colloid and Crystalloid Solutions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-0803
Record Dates: First submitted 2010-04-28; First posted 2010-05-05 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Plasma Volume Replacement; Surgery of the Pancreatic Head
Keywords: PVR; HES 130; pancreatic head; goal-directed; intraoperative PVR in elective surgery of the pancreatic head
MeSH Terms: interventions — HES 130-0.42-6:1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): hyper-oncotic colloid
  Interventions: Drug: HES 10%
- 2 (Active Comparator): iso-oncotic colloid
  Interventions: Drug: HES 6%
- 3 (Active Comparator): crystalloid
  Interventions: Drug: balanced electrolyte solution

INTERVENTIONS:
Drug: HES 10% — HES 10% dissolved in plasma adapted Ringer's solution (balanced solution).
  Arms: 1
Drug: HES 6% — HES 6% dissolved in plasma adapted Ringer's solution (balanced solution)
  Arms: 2
Drug: balanced electrolyte solution — plasma adapted Ringer's solution
  Arms: 3

SUMMARY:
The purpose of this study is to investigate the efficacy of target controlled fluid therapy with a hyper-oncotic balanced HES solution compared to an iso-oncotic HES solution in patients undergoing elective surgery of the pancreatic head. A third group receiving a balanced electrolyte solution (without colloidal volume replacement) will serve as a control for descriptive analysis.

ELIGIBILITY:
Inclusion:

* patients scheduled to undergo elective surgery of the pancreatic head
* patients who are willing to give of voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Institutional Ethics Committee (IEC) prior to all evaluations.

Exclusion:

* patients of American Society of Anesthesiologists (ASA) class > III
* heart failure defined as New York Heart Association (NYHA) class>2
* aneurysm of the ascending and thoracic aorta
* patients with Zenker's diverticle
* local oesophageal disease (oesophageal stricture, oesophageal varices, previous oesophageal surgery in past 6 months before study inclusion, pharyngeal pouch)
* patients receiving haemodialysis
* patients with known bleeding diatheses
* any bleeding disorder known from patient's history
* patients with a haematocrit <= 25% despite pre-operative transfusion
* renal insufficiency (serum creatinine > 130 µmol/l or >1.5 mg/dl) or oliguria or anuria
* impaired hepatic function defined as Mayo End-Stage Liver Disease (MELD) > 10 or liver cirrhosis Child-Pugh B or C
* additional contra-indications for investigational products

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
First endpoint: Intraoperatively required amount of HES (10%, 6%) (ml) | up to 8 hours
  Goal-directed (stroke volume) plasma volume therapy
Second endpoint: Time until fully on oral (solid) diet (days) | up to 15 days

SECONDARY OUTCOMES:
haemodynamics, arterial blood gas analysis, laboratory data, postoperative nausea and vomiting, adverse events, nursing delirium screening scale, several injury scores | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, Prof. Dr., Principal Investigator — Klinik für Anästhesie und operative Intensivmedizin, Charité-Universitätsmedizin Berlin, Campus Virchow-Klinikum
Locations (3):
- Germany (3):
  - Klinik für Anästhesie und operative Intensivmedizin, Charité-Universitätsmedizin Berlin, Berlin
  - Klinik für Anästhesie, operative Intensivmedizin und Schmerztherapie, Humboldt Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn